CLINICAL TRIAL: NCT05295732
Title: The ASCEND Study: A Phase III, Multicenter, Double Blinded Vehicle Controlled Study of TMB-001 - With a Parallel Optional Maximal Use Arm - in the Treatment of RXLI (X-linked) or ARCI Ichthyosis in Subjects Aged ≥6 Years
Brief Title: The ASCEND Study: Evaluating TMB-001 in the Treatment of RXLI or ARCI Ichthyosis
Acronym: ASCEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Timber Pharmaceuticals Inc. (Industry)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMB01-301; 2022-000459-35 (EudraCT Number)
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Ichthyosis
MeSH Terms: conditions — Ichthyosis

STUDY DESIGN:
Intervention Model Description: • Period 1 - Induction (3 weeks):
  At the beginning of the 3-week Induction Period, eligible subjects will be randomized (2:1 ratio) to either TMB-001 0.05% once-a-day (QD) or Vehicle QD treatment, with use of mandatory standardized bland emollient (Cetaphil™) provided by the Sponsor.
  • Period 2 - Treatment (9 weeks):
  The dosing frequency in the 9-week treatment period will be increased in each treatment group to TMB-001 0.05% BID or Vehicle BID. Mandatory bland emollient will be discontinued.
  • Period 3 - Maintenance (12 weeks):
  At Week 12, eligible subjects in the TMB-001 treatment group will be randomized (1:1 ratio) to an open-label treatment with TMB-001 0.05% BID or TMB-001 0.05% QD.
  Vehicle-treated subjects who achieved <1-point reduction in IGA score from Baseline are eligible to cross over to the TMB-001 0.05% BID treatment group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TMB-001 0.05% (Experimental): TMB-001 0.05% ointment: Induction phase QD for 3 weeks, followed by BID for 9 weeks. Maintenance therapy for additional 12 weeks randomized QD vs BID
  Interventions: Drug: TMB-001
- Vehicle (Placebo Comparator): Matching vehicle ointment: Induction phase QD for 3 weeks, followed by BID for 9 weeks. Cross over to 12 weeks TMB-001 0.05% BID.
  Interventions: Drug: Matching Vehicle
- Maximal use (Experimental): Optional Parallel Arm to evaluate the systemic exposure and safety of TMB-001 0.05% under conditions of maximal use.
  Interventions: Drug: TMB-001

INTERVENTIONS:
Drug: TMB-001 — Topical TMB-001 0.05% QD/BID
  Arms: Maximal use; TMB-001 0.05%
Drug: Matching Vehicle — Topical Vehicle
  Arms: Vehicle

SUMMARY:
This is a randomized, double-blind and vehicle-controlled Phase III study to evaluate the safety and efficacy of topical TMB-001 0.05% ointment for the treatment of congenital ichthyosis (CI) in subjects with either the RXLI or ARCI subtypes.

In addition, a subset of preselected centers will recruit subjects in parallel with either the RXLI or ARCI subtypes for enrollment into an Optional Maximal Use arm for evaluation of the systemic exposure and safety of topical TMB-001 0.05% ointment for the treatment of CI.

The Phase III Study is designed in three periods:

- Period 1 - Induction (3 weeks):

At the beginning of the 3-week Induction Period, eligible subjects will be randomized (2:1 ratio) to either TMB-001 0.05% once-a-day (QD) or Vehicle QD treatment, with use of mandatory standardized bland emollient (Cetaphil™) provided by the Sponsor.

- Period 2 - Treatment (9 weeks):

The dosing frequency in the 9-week treatment period will be increased in each treatment group to TMB-001 0.05% BID or Vehicle BID. Mandatory bland emollient will be discontinued.

- Period 3 - Maintenance (12 weeks):

At Week 12, eligible subjects in the TMB-001 treatment group will be randomized (1:1 ratio) to an open-label treatment with TMB-001 0.05% BID or TMB-001 0.05% QD. To be eligible, subjects must have achieved a ≥1-point reduction in IGA score from Baseline. Subjects with less than a 1-point reduction in IGA score from Baseline will be discontinued from the study.

Vehicle-treated subjects who achieved <1-point reduction in IGA score from Baseline are eligible to cross over to the TMB-001 0.05% BID treatment group. Subjects with a ≥1-point reduction in IGA score from Baseline on vehicle will be discontinued from the study.

Subjects at the end of the study or subjects discontinued from the study at any time will be followed-up for additional 2 weeks for AEs.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, vehicle-controlled Phase III study to evaluate the efficacy and safety of TMB-001 0.05% topical ointment in the treatment of CI. Subjects will be selected according to predefined entry criteria. The study treatment duration is 24 weeks and expected to be sufficient to show a treatment effect.

Isotretinoin is an approved active pharmacological ingredient with a long history of safe use in humans. However, isotretinoin is a known teratogen with an extremely high risk for severe birth defects if pregnancy occur while taking oral isotretinoin in any amount, even for a short period of time. Therefore oral, systemic isotretinoin requires an iPLEDGE program (iPLEDGE 2012), which is a risk management distribution program mandated by the FDA. To minimize pregnancy risks, women of childbearing potential (WOCBP) will only be enrolled if they agree to use highly effective methods of contraception consistently and correctly and undergo regular pregnancy testing.

To minimize bias, subjects will be blinded and randomly assigned to treatment with TMB-001 0.05% or Vehicle, additionally subjects who had previously been treated with TMB 001 will be excluded from this study but can be enrolled in the optional Maximal Use arm (in a subset of preselected centers). The use of a vehicle control group is consistent with FDA's standard for generating valid scientific evidence to definitively support safety and efficacy. The vehicle group accounts for the effects of treatment that do not depend on the test treatment. The study is designed to mitigate safety risks by using an initial 2:1 randomization (active treatment to vehicle), along with frequent clinic visits over the 12-week treatment period. The subsequent 1:1 randomization of eligible TMB-001 0.05% treated subjects to two dosing regimen (QD or BID) allows for assessment of the optimal TMB-001 0.05% maintenance therapy as well as provides additional safety data for 12 weeks. The cross-over of eligible subjects from the vehicle control group will also provide additional safety data.

Overall, the study design is considered to be scientifically robust and clinically relevant for evaluating TMB-001 0.05% treatment for the safe and effective treatment of CI.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 6 years of age and older at Visit 2 (Baseline).
2. Subject has provided written informed consent/assent. A subject under 18 years of age must provide written informed assent and be accompanied by the parent or legal guardian at the time of consent/assent signing. The parent or legal guardian must provide informed consent for the subject. If a subject becomes 18 years of age during the study, the subject must provide written informed consent at that time to continue study participation.
3. Females must be postmenopausal (defined as amenorrhea greater than 12 consecutive months in women 50 years of age and older), surgically sterile (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), or use 2 acceptable forms of birth control. WOCBP must have a negative serum pregnancy test at screening and negative urine pregnancy test (UPT) at Visit 2 (Baseline) (UPTs must have a minimum sensitivity to detect 25 mIU beta human chorionic gonadotropin [β hCG]/mL). Female subjects who become sexually active or begin to have relations with a partner during the study must agree to use 2 forms of birth control for 30 days prior to having relations and to continue such forms of birth control for the duration of the study.
4. Subject has clinical diagnosis of CI and has a genetic confirmation of either ARCI (including but not exclusively transglutaminase 1-deficient, ALOX-12B) or RXLI (e.g., deletion of steroid sulfatase gene) subtypes of CI. Other genetically confirmed ARCI-LI mutations can potentially be enrolled as long as the phenotype is consistent with ARCI and the other inclusion criteria are met, as determined by the Investigator.
5. The amount of CI affected skin in the Treatment Area at Baseline will be between a minimum of 10% and maximum of 90% of the total BSA (1% BSA is approximately equal to the surface area of the subject's palm and fingers, with the fingers extended yet grouped together, creating a flat oval-like surface area).

   • For the Optional Maximal Use arm: The amount of CI affected skin in the Treatment Area at Baseline will be between a minimum of 75% and maximum of 90% of the total BSA.
6. Documented history of moderate to severe disease at Screening. Subject's designated VIIS Assessment Areas at Baseline (not applicable for Optional Maximal Use arm):

   * Include any of the 4 VIIS Assessment Areas that have some CI disease involving: (a) the upper back from the posterior axillary fold to the other encompassing the T1-T10, (b) the upper arm (excluding elbows), left or right, (c) the shin/lower leg (the portion below the proximal aspect of the kneecap), left or right, and (d) dorsal foot (left or right); AND
   * At least 2 of the 4 VIIS Assessment Areas MUST have a scaling score of 3 or more.
7. Subject's IGA score in the Treatment Area at Baseline must be 3 or more.
8. Subject and parent/guardian (if applicable) are willing and able to apply the study treatment(s) as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
9. Subject, in the Investigator's opinion, is in good general health and free of any disease state or physical condition that might impair evaluation of the Treatment Areas or exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has inflammatory skin diseases that confound the interpretation of results (e.g., atopic dermatitis) unrelated to ichthyosis.
3. Subject has genetic abnormality consistent with non-lamellar type or syndromic ichthyoses (including but not exclusively KRT1, KRT10, KRT2, GJB3, GJB4, CDSN)
4. Subject, in the Treatment Areas, has used: (a) any topical prescription or over-the-counter (OTC) therapies (except emollients, keratolytics, and topical steroids - see below), that are intended for, or that in the opinion of the Investigator, may improve CI within 2 weeks of Visit 2 (Baseline), or (b) keratolytics or topical corticosteroids within 5 days prior to Visit 2 (Baseline).
5. Subject, in the Treatment Areas, has used TMB-001 in the past or oral isotretinoin in the past 12 months (not applicable for Optional Maximal Use arm).
6. Subject has used any topical products in the Treatment Areas, including bland emollients, on Visit 2 (Baseline).
7. Subject has used ultraviolet (UV) treatment within 4 weeks prior to Visit 2 (Baseline).
8. Subject has undergone systemic therapies using vitamin A supplements or St. John's Wort within 4 weeks prior to Visit 2 (Baseline). Note: Use of a multivitamin including vitamin A is not exclusionary provided it is taken as directed on the packaging.
9. Subject is immunosuppressed (e.g., human immunodeficiency virus, systemic malignancy, graft host disease) or receives systemic immunotherapy.
10. Subject is currently taking concomitant immunosuppressive drugs, including systemic corticosteroids, within 2 weeks of Visit 2 (Baseline).
11. Subject has untreated secondary infections; however, subject may become eligible after successful treatment of his/her infection(s) at the Investigator's discretion.
12. Subject is currently enrolled in an investigational drug or device study or has used an investigational drug or investigational device treatment within 30 days or five half-lives prior to Visit 2 (Baseline).
13. Subject has lesions suspicious for skin cancer (if skin cancer is not ruled out by biopsy) or untreated skin cancers within the Treatment Areas.
14. Subject has a physical condition or other dermatologic disorder that, in the Investigator's opinion, might impair evaluation of CI, or that exposes the subject to unacceptable risk by study participation.
15. Subjects with ALT or AST >2 x Upper Limit of Normal (ULN) and/or creatinine >1.5 x ULN.
16. Subject is unable to communicate or cooperate with the Investigator due to language problems, impaired cerebral function, or physical limitations.
17. Subject has a history of drug or alcohol abuse within the past 6 months, or if suspected to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the Investigator.
18. Subject has a history of sensitivity to any of the ingredients in the study treatments.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (18):
  - U.S. Dermatology Partners, Phoenix, Arizona
  - Stanford University School of Medicine, Palo Alto, California
  - About Skin Dermatology, Centennial, Colorado
  - Yale Center for Clinical Investigation, New Haven, Connecticut
  - Department of Dermatology and Cutaneous Surgery, University of Miami, Miami, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Associated Skincare Specialists, New Brighton, Minnesota
  - University of Mississippi Medical Center (UMMC), Jackson, Mississippi
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Optima Research, Boardman, Ohio
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Austin Institute for Clinical Research, Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Virginia Clinical Research-Pariser Dermatology Specialists, Norfolk, Virginia
  - North Sound Dermatology, Mill Creek, Washington
- Canada (4):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SickKids Hospital, Toronto, Ontario
- France (4):
  - Hôpital Femme Mère Enfant, Bron
  - CHU de Nantes Hotel Dieu, Nantes
  - Hopital Necker APHP, Paris
  - Hopital Larrey CHU Toulouse, Toulouse
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Katholisches Kinderkrankenhaus Wilhelmstift GmbH, Hamburg
  - Münster University Hospital, Münster
- Italy (5):
  - U.O. di Dermatologia e Venereologia Universitaria, Bari
  - U.O. di Dermatologia Dipartimento di Medicina Specialistica, Diagnostica e Sperimentale, Bologna
  - Ambulatorio di Malattie Rare Dermatologiche e Immunopatologia Cutanea, Florence
  - Fondazione IRCCS Ospedale Maggiore Policlinico Milano, Area Materno Infantile - SC pediatria Pneumoinfettivologia, Milan
  - U.O.C. di Dermatologia Dipartimento Pediatrico Universitario Ospedaliero, Roma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 34 sites across the United States, Canada, Germany, France, and Italy enrolled subjects, and 33 of these sites randomized subjects.
Groups:
- TMB-001 0.05%: In the first 3 weeks of the 12-week double-blind primary dosing period, subjects were randomized to TMB-001 0.05% QD with use of mandatory standardized bland emollient (Cetaphil™). For the last 9 weeks of the 12 week double-blind primary dosing period, the subjects continued with TMB-001 0.05% at the increased dosing frequency of BID. Mandatory bland emollient was discontinued.
- Vehicle: In the first 3 weeks of the 12-week double-blind primary dosing period, subjects were randomized to Vehicle QD treatment, with use of mandatory standardized bland emollient (Cetaphil™). For the last 9 weeks of the 12-week double-blind primary dosing period, the subjects continued with Vehicle at the increased dosing frequency of BID. Mandatory bland emollient was discontinued.
- TMB-001 0.05% QD: At Week 12, TMB-001 0.05% BID treatment responders (who had achieved a ≥1-point reduction in IGA score from baseline) were re-randomized (1:1 ratio) to 12 weeks of open-label treatment with TMB-001 0.05% BID or TMB-001 0.05% QD. Subjects with less than a 1-point reduction in IGA score from baseline were discontinued from the study. Vehicle-treated subjects who achieved <1-point reduction in IGA score from baseline by week 12, were eligible to cross over to 12 weeks of open-label treatment with TMB-001 0.05% BID treatment. Subjects with a ≥1-point reduction in IGA score from baseline on vehicle were discontinued from the study.
- TMB-001 0.05% BID: At Week 12, TMB-001 0.05% BID treatment responders (who had achieved a ≥1-point reduction in IGA score from baseline) were re-randomized (1:1 ratio) to 12 weeks of open-label treatment with TMB-001> 0.05% BID or TMB-001 0.05% QD. Subjects with less than a 1-point reduction in IGA score from baseline were discontinued from the study. Vehicle-treated subjects who achieved <1-point reduction in IGA score from baseline by week 12, were eligible to cross over to 12 weeks of open-label treatment with TMB-001 0.05% BID treatment. Subjects with a ≥1-point reduction in IGA score from baseline on vehicle were discontinued from the study.
- Maximal Use: The optional maximal use arm part of the trial was conducted under the same protocol number for operational reasons, but with separate design, objective, and patients. Adult and pediatric subjects, at a subset of preselected centers, were enrolled in an open-label Optional Maximal Use Arm to evaluate the systemic exposure and safety of TMB-001 0.05% for the treatment of congenital ichthyosis under maximal use conditions. Initially, adult and pediatric subjects with congenital ichthyosis were dosed for 14 days with TMB-001 0.05% BID. Following an interim pharmacokinetic (PK) analysis and based on the exposure data for subjects aged ≥12 years, pediatric subjects aged 6 to 11 years began dosing with TMB-001 0.05% BID for 14> days. Following the 14-day PK assessment period, subjects received TMB-001 0.05% BID treatment for 10 weeks to provide additional safety and limited efficacy data.
Period: Phase 3: Double-blind / MUsT: Treatment
Arm/Group | TMB-001 0.05% | Vehicle | TMB-001 0.05% QD | TMB-001 0.05% BID | Maximal Use
Started | 79 | 40 | 0 | 0 | 34
Dosed | 78 | 38 | 0 | 0 | 34
Completed | 65 | 36 | 0 | 0 | 32
Not Completed | 14 | 4 | 0 | 0 | 2
Not completed — Various reasons | 14 | 4 | 0 | 0 | 2
Period: Phase 3: Open-label / MUsT: Maintenance
Arm/Group | TMB-001 0.05% | Vehicle | TMB-001 0.05% QD | TMB-001 0.05% BID | Maximal Use
Started | 0 | 0 | 28 | 38 | 32
Completed | 0 | 0 | 28 | 37 | 31
Not Completed | 0 | 0 | 0 | 1 | 1
Not completed — Various reasons | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: TMB-001 0.05% and vehicle: Intent-to-Treat (ITT) population = all randomized subjects who received at least one dose of study medication. > Maximal Use = all subjects enrolled in the maximal use arm who receive at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | TMB-001 0.05% | Vehicle | Maximal Use | Total
Number analyzed (Participants) | 78 | 38 | 34 | 150
Age, Customized [Count of Participants; unit: Participants]
  Age: 6-11 years | 16 | 8 | 9 | 33
  Age: 12-16 years | 19 | 8 | 7 | 34
  Age: >=17 years | 43 | 22 | 18 | 83
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 15 | 16 | 60
  Male | 49 | 23 | 18 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 28 | 19 | 25 | 72
  Unknown or Not Reported | 48 | 17 | 7 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 2 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 2 | 5 | 7 | 14
  White | 57 | 25 | 21 | 103
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 16 | 5 | 2 | 23
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.903 (5.4218) | 24.092 (7.6000) | 24.468 (8.6960) | 23.559 (6.8388)

OUTCOME MEASURES:

1. Primary Outcome: Change in Investigator Global Assessment (IGA) Score
Description: Comparison of proportions of subjects in percentages with ≥2-point changes from Baseline in Investigator Global Assessment (IGA)-scaling and fissuring scores in the Treatment Area at Week 12 between TMB-001 0.05% and vehicle-treated subjects. Investigator's Global Assessment Score is a 0-4 scale, where 0 is clear and 4 is severe.
Time Frame: 12 weeks
Population: For the primary efficacy endpoint, missing Week 12 IGA scores were imputed by a multiple imputation approach and IGA responder status was derived from the imputed values. The analysis was then performed on each of the 50 imputed datasets. The final proportion of responders is the average proportion across all 50 imputed datasets hence the proportion is not an exact fraction of the total number of subjects.
Measure: Number; unit: percentage of responders
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 78 | 38
percentage of responders | 41.4 | 44.9
Statistical Analysis 1: Comparison: TMB-001 0.05% vs Vehicle; Test type: Superiority; p = 0.39, Cochran-Mantel-Haenszel; treatment difference = -1.0, 95% CI 2-sided [-18.4 to 16.5]

2. Secondary Outcome: Number of Subjects With IGA Scores
Description: Comparison of proportion of subjects in percentages with IGA scores of clear or almost clear at Week 12 between TMB-001 0.05% and vehicle-treated subjects. Investigator's Global Assessment Score is a 0-4 scale, where 0 is clear and 4 is severe.
Time Frame: 12 weeks
Population: Missing values were imputed by a multiple imputation approach and the final proportion of responders is the average proportion across all imputed datasets, hence the proportion is not an exact fraction of the total number of subjects.
Measure: Number; unit: percentage of responders
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 78 | 38
percentage of responders | 35.8 | 38.9

3. Secondary Outcome: Change in IGA-scaling Severity Sub-score
Description: Comparison of proportion of subjects in percentages who achieve IGA-scaling severity sub-score improvement ≥ 2-points from Baseline to Week 12 between TMB-001 0.05% and vehicle-treated subjects. Investigator's Global Assessment Score is a 0-4 scale, where 0 is clear and 4 is severe.
Time Frame: 12 weeks
Population: Data is not available for 3 participants in the TMB-001 0.05% group and for 2 participants in the vehicle group. Missing values were imputed by a multiple imputation approach and the final proportion of responders is the average proportion across all imputed datasets, hence the proportion is not an exact fraction of the total number of subjects.
Measure: Number; unit: percentage of responders
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 75 | 36
percentage of responders | 40.4 | 36.4

4. Secondary Outcome: Change in Worst Itch-Quality of Life (QoL) Scores
Description: Comparison of proportion of subjects in percentages with ≥4-point improvement from baseline in Worst Itch-QoL scores at Week 12 in subjects with baseline WI-NRS of ≥7 between TMB-001 0.05% and vehicle-treated subjects. Itch-Numeric Rating Scale (I-NRS) and Worst Itch-Numeric Rating Scale (WI-NRS) is an 0-10 scale where 0 is "no itching" and 10 is "worst itch imaginable".
Time Frame: 12 weeks
Population: Data is not available for 59 participants in the TMB-001 0.05% group and for 29 participants in the vehicle group. Missing values were imputed by a multiple imputation approach and the final proportion of responders is the average proportion across all imputed datasets, hence the proportion is not an exact fraction of the total number of subjects.
Measure: Number; unit: percentage of responders
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 19 | 9
percentage of responders | 54.4 | 68.7

5. Secondary Outcome: Change in Visual Index of Ichthyosis Severity (VIIS) Score
Description: Comparison of proportion of subjects in percentages who achieve 50% reduction from Baseline in VIIS-scaling scores at Week 12 in all areas with Baseline VIIS score ≥3 between TMB-001 0.05% and vehicle-treated subjects. Visual Index for Ichthyosis Severity Score is a 0-4 scale where 0 is clear and 4 is severe.
Time Frame: 12 weeks
Population: Data is not available for 4 participants in the TMB-001 0.05% group. Missing values were imputed by a multiple imputation approach and the final proportion of responders is the average proportion across all imputed datasets, hence the proportion is not an exact fraction of the total number of subjects.
Measure: Number; unit: percentage of responders
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 74 | 38
percentage of responders | 47.2 | 42.7

6. Secondary Outcome: Change in VIIS Score
Description: Comparison of proportion of subjects in percentages who achieve 25% reduction from Baseline in VIIS-scaling scores at Week 12 in all areas with Baseline VIIS score ≥3 between TMB-001 0.05% and vehicle-treated subjects. Visual Index for Ichthyosis Severity Score is a 0-4 scale where 0 is clear and 4 is severe.
Time Frame: 12 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of responders
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 74 | 38
percentage of responders | 71.3 | 64.1

7. Secondary Outcome: Change in IGA-fissuring Severity Sub-scores
Description: Comparison of proportion of subjects in percentages achieving ≥2 point improvement in IGA-fissuring severity sub-scores from Baseline to Week 12 between TMB-001 0.05% and vehicle-treated subjects. Investigator's Global Assessment Score is a 0-4 scale, where 0 is clear and 4 is severe.
Time Frame: 12 weeks
Population: Data is not available for 48 participants in the TMB-001 0.05% group and for 21 participants in the vehicle group. Missing values were imputed by a multiple imputation approach and the final proportion of responders is the average proportion across all imputed datasets, hence the proportion is not an exact fraction of the total number of subjects.
Measure: Number; unit: percentage of responders
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 30 | 17
percentage of responders | 54.1 | 57.9

8. Secondary Outcome: Change in IGA Score
Description: Comparison of proportions of subjects in percentages achieving ≥2-point improvement from Baseline in IGA scores at Week 24 between subjects randomized to TMB-001 0.05% BID and QD maintenance dosing. Investigator's Global Assessment Score is a 0-4 scale, where 0 is clear and 4 is severe.
Time Frame: 24 weeks
Population: Data reported for the re-randomized TMB-001 0.05% responders subjects in TMB-001 0.05% BID group. Missing values were imputed by a multiple imputation approach and the final proportion of responders is the average proportion across all imputed datasets, hence the proportion is not an exact fraction of the total number of subjects.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- TMB-001 0.05% QD: At Week 12, TMB-001 0.05% BID treatment responders (who had achieved a ≥1-point reduction in IGA score from baseline) were re-randomized (1:1 ratio) to 12 weeks of open-label treatment with TMB-001> 0.05% BID or TMB-001 0.05% QD. Subjects with less than a 1-point reduction in IGA score from baseline were discontinued from the study. Vehicle-treated subjects who achieved <1-point reduction in IGA score from baseline by week 12, were eligible to cross over to 12 weeks of open-label treatment> with TMB-001 0.05% BID treatment. Subjects with a ≥1-point reduction in IGA score from baseline on vehicle were> discontinued from the study.
- TMB-001 0.05% BID: At Week 12, TMB-001 0.05% BID treatment responders (who had achieved a ≥1-point reduction in IGA score from baseline) were re-randomized (1:1 ratio) to 12 weeks of open-label treatment with TMB-001 0.05% BID or TMB-001 0.05% QD. Subjects with less than a 1-point reduction in IGA score from baseline were discontinued from the study. Vehicle-treated subjects who achieved <1-point reduction in IGA score from baseline by week 12, were eligible to cross over to 12 weeks of open-label treatment with TMB-001 0.05% BID treatment. Subjects with a ≥1-point reduction in IGA score from baseline on vehicle were discontinued from the study.
Arm/Group | TMB-001 0.05% QD | TMB-001 0.05% BID
Number analyzed (Participants) | 28 | 27
percentage of responders | 57.1 [38.8 to 75.5] | 85.2 [71.8 to 98.6]

9. Secondary Outcome: Change in VIIS Score
Description: Comparison of proportion of subjects in percentages who achieve 50% reduction from Baseline in VIIS-scaling scores at Week 24 in all areas with Baseline VIIS score ≥3 between subjects randomized to TMB-001 0.05% BID and QD maintenance dosing. Visual Index for Ichthyosis Severity Score is a 0-4 scale where 0 is clear and 4 is severe.
Time Frame: 24 weeks
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | TMB-001 0.05% QD | TMB-001 0.05% BID
Number analyzed (Participants) | 28 | 27
percentage of responders | 63.0 [44.7 to 81.2] | 85.2 [71.8 to 98.6]

10. Secondary Outcome: Change in Ichthyosis Quality of Life (IQoL)-32 Scores
Description: Comparison of proportions of subjects in percentages with ≥11-point changes from Baseline in IQOL-32 scores at Week 12 between TMB-001 0.05% and vehicle-treated subjects. The IQoL-32 is a questionnaire containing 32, each scored from 0 to 4 ('not applicable', 'not at all', 'a little', 'a lot', 'tremendously') for a total score that varies between 0 and 128. A higher score, the higher impact on quality of life.
Time Frame: 12 weeks
Population: Data is not available for 44 participants in the TMB-001 0.05% group and for 17 participants in the vehicle group.
Measure: Number; unit: percentage of responders
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 34 | 21
percentage of responders | 47.1 | 9.5

11. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) Scores
Description: Comparison of proportion of subjects in percentages with reduction from Baseline in DLQI ≥4 points at Week 12 between TMB-001 0.05% and vehicle-treated subjects in adult subjects with Baseline scores ≥11. The age-appropriate questionnaire contains 10 questions scored from 0 (no impact of skin disease on QoL) to 30 (maximum impact on QoL).
Time Frame: 12 weeks
Population: Data is not available for 63 participants in the TMB-001 0.05% group and for 30 participants in the vehicle group.
Measure: Number; unit: percentage of responders
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 15 | 8
percentage of responders | 86.7 | 37.5

12. Secondary Outcome: Change in Children's Dermatology Life Quality Index (CDLQI) Scores
Description: Comparison of proportion of pediatric subjects in percentages with reduction from Baseline in CDLQI ≥4 points at Week 12 between TMB-001 0.05% and vehicle-treated subjects in pediatric subjects with Baseline scores of ≥13. The age-appropriate questionnaire contains 10 questions scored from 0 (no impact of skin disease on QoL) to 30 (maximum impact on QoL).
Time Frame: 12 weeks
Population: Only 5 pediatric subjects had Baseline scores of ≥13 in the TMB-001 0.05% group. No pediatric subjects had Baseline scores of ≥13 in the vehicle group.
Measure: Number; unit: percentage of responders
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 5 | 0
percentage of responders | 80.0 |

13. Secondary Outcome: Change in Itch-Quality of Life Scores - I-NRS
Description: Comparison of proportions of subjects in percentages with I-NRS improvement ≥4 points from Baseline in Itch-QoL scores (in subjects with Baseline I-NRS ≥7) at Week 24 between subjects randomized to TMB-001 0.05% BID and QD maintenance dosing.
Time Frame: 24 weeks
Population: No participants in the TMB-001 0.05% QD Group had Baseline I-NRS scores ≥7 and therefore, 0 participants in this Group were analyzed for this measure. Data is not available for 37 participants in the TMB-001 0.05% BID group.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- TMB-001 0.05% QD; TMB-001 0.05% BID: At Week 12, TMB-001 0.05% BID treatment responders (who had achieved a ≥1-point reduction in IGA score from baseline) were re-randomized (1:1 ratio) to 12 weeks of open-label treatment with TMB-001 0.05% BID or TMB-001 0.05% QD. Subjects with less than a 1-point reduction in IGA score from baseline were discontinued from the study. Vehicle-treated subjects who achieved <1-point reduction in IGA score from baseline by week 12, were eligible to cross over to 12 weeks of open-label treatment with TMB-001 0.05% BID treatment. Subjects with a ≥1-point reduction in IGA score from baseline were discontinued from the study.
Arm/Group | TMB-001 0.05% QD | TMB-001 0.05% BID
Number analyzed (Participants) | 0 | 1
percentage of responders |  | 100 [100.0 to 100.0]

14. Secondary Outcome: Change in Itch-Quality of Life Scores - WI-NRS
Description: Comparison of proportions of subjects in percentages with WI-NRS improvement ≥4 points from Baseline in Itch-QoL scores (in subjects with Baseline WI-NRS ≥7) at Week 24 between subjects randomized to TMB-001 0.05% BID and QD maintenance dosing.
Time Frame: 24 weeks
Population: Data is not available for 25 participants in the TMB-001 0.05% QD group and for 23 participants in the TMB-001 0.05% BID group. In addition, 11 participants in the TMB-001 0.05% BID group randomized to vehicle in the double-blinded period were not included. Missing values were imputed by a multiple imputation approach and the final proportion of responders is the average proportion across all imputed datasets, hence the proportion is not an exact fraction of the total number of subjects.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | TMB-001 0.05% QD | TMB-001 0.05% BID
Number analyzed (Participants) | 3 | 4
percentage of responders | 66.7 [0.00 to 100.0] | 75.0 [19.2 to 100.0]

15. Secondary Outcome: Change in DLQI Scores
Description: Comparison of proportions of adult subjects in percentages with DLQI changes of ≥4-point from Baseline scores (in subjects with Baseline scores ≥11) at Week 24 randomized to TMB-001 0.05% BID and QD maintenance dosing. The age-appropriate questionnaire contains 10 questions scored from 0 (no impact of skin disease on QoL) to 30 (maximum impact on QoL).
Time Frame: 24 weeks
Population: Data is not available for 24 participants in the TMB-001 0.05% QD group and for 23 participants in the TMB-001 0.05% BID group. In addition, 11 participants in the TMB-001 0.05% BID group randomized to vehicle in the double-blinded period were not included.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | TMB-001 0.05% QD | TMB-001 0.05% BID
Number analyzed (Participants) | 4 | 4
percentage of responders | 75.0 [32.6 to 100.0] | 100 [100.0 to 100.0]

16. Secondary Outcome: Change in CDLQI Scores
Description: Comparison of proportions of pediatric subjects in percentages with CDLQI changes of ≥4-point from Baseline scores (in subjects with Baseline scores ≥13) at Week 24 randomized to TMB-001 0.05% BID and QD maintenance dosing. The age-appropriate questionnaire contains 10 questions scored from 0 (no impact of skin disease on QoL) to 30 (maximum impact on QoL).
Time Frame: 24 weeks
Population: Only 1 pediatric subjects had Baseline scores of ≥13 in the TMB-001 0.05% QD group, and 3 pediatric subjects had Baseline scores of ≥13 in the TMB-001 0.05% BID group.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- TMB-001 0.05% BID: At Week 12, TMB-001 0.05% BID treatment responders (who had achieved a ≥1-point reduction in IGA score from baseline) were re-randomized (1:1 ratio) to 12 weeks of open-label treatment with TMB-001 0.05% BID or TMB-001 0.05% QD. Subjects with less than a 1-point reduction in IGA score from baseline on vehicle were discontinued from the study. Vehicle-treated subjects who achieved <1-point reduction in IGA score from baseline by week 12, were eligible to cross over to 12 weeks of open-label treatment with TMB-001 0.05% BID treatment. Subjects with a ≥1-point reduction in IGA score from baseline were discontinued from the study.
Arm/Group | TMB-001 0.05% QD | TMB-001 0.05% BID
Number analyzed (Participants) | 1 | 3
percentage of responders | 100 [100.0 to 100.0] | 100 [100.0 to 100.0]

17. Secondary Outcome: Change in IQoL-32 Scores
Description: Proportions of subjects in percentages with ≥11-point change from Baseline in IQoL-32 at Week 24 between subjects randomized to TMB-001 0.05% BID and QD maintenance dosing in adult subjects. The IQoL-32 is a questionnaire containing 32, each scored from 0 to 4 ('not applicable', 'not at all', 'a little', 'a lot', 'tremendously') for a total score that varies between 0 and 128. A higher score, the higher impact on quality of life.
Time Frame: 24 weeks
Population: Data is not available for 18 participants in the TMB-001 0.05% QD group and for 17 participants in the TMB-001 0.05% BID group. In addition, 11 participants in the TMB-001 0.05% BID group randomized to vehicle in the double-blinded period were not included.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- TMB-001 0.05% QD; TMB-001 0.05% BID: At Week 12, TMB-001 0.05% BID treatment responders (who had achieved a ≥1-point reduction in IGA score from baseline) were re-randomized (1:1 ratio) to 12 weeks of open-label treatment with TMB-001 0.05% BID or TMB-001 0.05% QD. Subjects with less than a 1-point reduction in IGA score from baseline on vehicle were discontinued from the study. Vehicle-treated subjects who achieved <1-point reduction in IGA score from baseline by week 12, were eligible to cross over to 12 weeks of open-label treatment with TMB-001 0.05% BID treatment. Subjects with a ≥1-point reduction in IGA score from baseline were discontinued from the study.
Arm/Group | TMB-001 0.05% QD | TMB-001 0.05% BID
Number analyzed (Participants) | 10 | 10
percentage of responders | 40.0 [9.6 to 70.4] | 60.0 [29.6 to 90.4]

18. Secondary Outcome: To Investigate the Proportion of Subjects Experiencing Local Skin Reactions (LSRs) With Topically Applied TMB-001 0.05% Ointment.
Description: Comparison of proportion of subjects in percentages experiencing LSRs through Week 12 between TMB-001 0.05% and vehicle-treated subjects.
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 78 | 38
percentage of participants | 64.1 [52.4 to 74.7] | 36.8 [21.8 to 54.0]

19. Secondary Outcome: To Investigate the Proportion of Subjects Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: Comparison of proportion of subjects in percentages experiencing TEAEs through Week 12 between TMB-001 0.05% and vehicle-treated subjects.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 78 | 38
percentage of participants | 76.9 | 63.2

20. Secondary Outcome: To Investigate the Proportion of Subjects Experiencing LSRs With Topically Applied TMB-001 0.05% Ointment.
Description: Comparison of proportion of subjects in percentages experiencing LSRs through Week 24 between subjects randomized to TMB-001 0.05% BID and QD maintenance dosing.
Time Frame: 24 weeks
Population: Data reported for the re-randomized TMB-001 0.05% responders subjects in TMB-001 0.05% BID group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TMB-001 0.05% QD | TMB-001 0.05% BID
Number analyzed (Participants) | 28 | 27
percentage of participants | 32.1 [15.9 to 52.4] | 40.7 [22.4 to 61.2]

21. Secondary Outcome: To Investigate the Proportion of Subjects Experiencing TEAEs
Description: Comparison of proportion of subjects in percentages experiencing TEAEs through Week 24.
Time Frame: 24 weeks
Population: Data reported for the re-randomized TMB-001 0.05% responders subjects in TMB-001 0.05% BID group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TMB-001 0.05% QD | TMB-001 0.05% BID
Number analyzed (Participants) | 28 | 27
percentage of participants | 53.6 [33.9 to 72.5] | 48.1 [28.7 to 68.1]

22. Secondary Outcome: To Investigate the Proportion of Subjects Demonstrating Clinically Confirmed Allergic Contact Dermatitis
Description: Comparison of proportion of subjects in percentages demonstrating clinically confirmed allergic contact dermatitis by patch testing through Week 12 between TMB-001 0.05% and vehicle-treated subjects.
Time Frame: Through week 12
Measure: Number; unit: percentage of participants
Arm/Group | TMB-001 0.05% | Vehicle
Number analyzed (Participants) | 78 | 38
percentage of participants | 0 | 0

23. Secondary Outcome: Maximal Use Arm: Isotretinoin, Tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin - Cmax After Multiple Dosing - Adults
Description: maximal observed plasma concentration.
  > Assessment of concentrations of isotretinoin, tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin.
Time Frame: 14 days
Population: Data is not available for 24 participants in the Maximal use group.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Maximal Use: The optional maximal use arm part of the trial was conducted under the same protocol number for operational reasons, but with separate design, objective, and patients. Adult and pediatric subjects, at a subset of preselected centers, were enrolled in an open-label Optional Maximal Use Arm to evaluate the systemic exposure and safety of TMB-001 0.05% for the treatment of congenital ichthyosis under maximal use conditions. Initially, adult and pediatric subjects with congenital ichthyosis were dosed for 14 days with TMB-001 0.05% BID. Following an interim pharmacokinetic (PK) analysis and based on the exposure data for subjects aged ≥12 years, pediatric subjects aged 6 to 11 years began dosing with TMB-001 0.05% BID for 14
  > days. Following the 14-day PK assessment period, subjects received TMB-001 0.05% BID treatment for 10 weeks to provide additional safety and limited efficacy data.
Arm/Group | Maximal Use
Number analyzed (Participants) | 10
ng/mL
  Isotretinoin | 4.13 (6.48)
  4-Oxo-Isotretinoin | 16.7 (26)
  Tretinoin | 0.04 (0.12)
  4-oxo-tretinoin | 0.00 (0.00)

24. Secondary Outcome: Maximal Use Arm: Isotretinoin, Tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin - Cmax After Multiple Dosing - Adolescents
Description: as for outcome 23
Time Frame: 14 days
Population: Data is not available for 32 participants in the Maximal use group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Maximal Use
Number analyzed (Participants) | 2
ng/mL
  Isotretinoin | 7.7 (1.17)
  4-Oxo-Isotretinoin | 25.44 (10.11)
  Tretinoin | 4.52 (6.39)
  4-oxo-tretinoin | 3.60 (5.08)

25. Secondary Outcome: Maximal Use Arm: Isotretinoin, Tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin - AUC0-24 After Multiple Dosing - Adults
Description: AUC0-24 = area under the curve over the first 24 hours post dose.
  > Assessment of concentrations of isotretinoin, tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin.
Time Frame: 0-24hrs after dose
Population: Data is not available for 24 participants in the Maximal use group.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Maximal Use
Number analyzed (Participants) | 10
hr*ng/mL
  Isotretinoin | 78.44 (122.08)
  4-Oxo-Isotretinoin | 352.95 (577.05)
  Tretinoin | 0.17 (0.54)
  4-oxo-tretinoin | 0.00 (0.00)

26. Secondary Outcome: Maximal Use Arm: Isotretinoin, Tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin - AUC0-24 After Multiple Dosing - Adolescents
Description: as for outcome 25
Time Frame: 0-24hrs after dose
Population: Data is not available for 32 participants in the Maximal use group.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Maximal Use
Number analyzed (Participants) | 2
hr*ng/mL
  Isotretinoin | 101.34 (61.15)
  4-Oxo-Isotretinoin | 432.96 (121.81)
  Tretinoin | 13.74 (19.43)
  4-oxo-tretinoin | 10.15 (14.35)

27. Secondary Outcome: Maximal Use Arm: Isotretinoin, Tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin - Tmax After Multiple Dosing - Adults
Description: Tmax = time to maximal plasma concentration.
  > Assessment of concentrations of isotretinoin, tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin.
Time Frame: 14 days
Population: Data is not available for 24 participants in the Maximal use group.
Measure: Median (Full Range); unit: hours
Arm/Group | Maximal Use
Number analyzed (Participants) | 10
hours
  Isotretinoin | 1.50 [0 to 24]
  4-Oxo-Isotretinoin | 5 [0 to 24]
  Tretinoin | 0.00 [0.00 to 6.00]
  4-oxo-tretinoin | 0.00 [0.00 to 0.00]

28. Secondary Outcome: Maximal Use Arm: Isotretinoin, Tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin - Tmax After Multiple Dosing - Adolescents
Description: as for outcome 27
Time Frame: 14 days
Population: Data is not available for 32 participants in the Maximal use group.
Measure: Median (Full Range); unit: hours
Arm/Group | Maximal Use
Number analyzed (Participants) | 2
hours
  Isotretinoin | 14 [4 to 24]
  4-Oxo-Isotretinoin | 18 [12 to 24]
  Tretinoin | 2.00 [0.00 to 4.00]
  4-oxo-tretinoin | 1.00 [0.00 to 2.00]

29. Secondary Outcome: Maximal Use Arm: Isotretinoin, Tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin - Steady State Concentration After Multiple Dosing - Children
Description: Assessment of concentrations of isotretinoin, tretinoin, 4-oxo-tretinoin and 4-oxo-isotretinoin.
Time Frame: 14 days
Population: Data is not available for 27 participants in the Maximal use group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Maximal Use
Number analyzed (Participants) | 7
ng/mL
  Isotretinoin | 1.27 (1.2)
  4-Oxo-Isotretinoin | 9.53 (6.13)
  Tretinoin | 0 (0)
  4-oxo-tretinoin | 0 (0)

30. Secondary Outcome: Maximal Use Arm: Safety and Tolerability - LSRs
Description: Local skin reactions (burnings/stinging, erythema, erosions and edema) are reported as LSRs.
Time Frame: 12 weeks
Measure: Number; unit: events
Arm/Group | Maximal Use
Number analyzed (Participants) | 34
events
  Erythema | 16
  Erosions | 7
  Edema | 2
  Burning/stinging | 17

31. Secondary Outcome: Maximal Use Arm: Safety and Tolerability - TEAEs
Description: Local safety are reported as severe TEAEs related to treatment area.
Time Frame: 12 weeks
Measure: Number; unit: events
Arm/Group | Maximal Use
Number analyzed (Participants) | 34
events
  Pruritus | 2
  Administration site reactions | 8

ADVERSE EVENTS:
Time Frame: 24 weeks for the phase 3 trial part and 12 weeks for the Maximal use arm
Description: TEAEs. An AE is defined as treatment emergent if the AE start on or after treatment start until 30 days after treatment end date.
Groups:
- Double-blinded Phase: TMB-001 0.05%: Double-blinded phase: TMB-001 0.05% (N=78)
- Double-blinded Phase: Vehicle: Double-blinded phase: Vehicle (N=38)
- Open-label Phase: TMB-001 0.05% QD: Open-label phase: TMB-001 0.05% QD (N=28)
- Open-label Phase: TMB-001 0.05% BID: Open-label phase: TMB-001 0.05% BID (N=38)
- Maximal Use: Maximal use (N=34)
Arm/Group | Double-blinded Phase: TMB-001 0.05% | Double-blinded Phase: Vehicle | Open-label Phase: TMB-001 0.05% QD | Open-label Phase: TMB-001 0.05% BID | Maximal Use
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/38 | 0/28 | 0/38 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/78 | 0/38 | 0/28 | 0/38 | 0/34
Other Adverse Events (participants affected / at risk) | 47/78 | 17/38 | 11/28 | 14/38 | 22/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blinded Phase: TMB-001 0.05% (N=78) | Double-blinded Phase: Vehicle (N=38) | Open-label Phase: TMB-001 0.05% QD (N=28) | Open-label Phase: TMB-001 0.05% BID (N=38) | Maximal Use (N=34)
Viral rash (Infections and infestations) | 1 (1) | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blinded Phase: TMB-001 0.05% (N=78) | Double-blinded Phase: Vehicle (N=38) | Open-label Phase: TMB-001 0.05% QD (N=28) | Open-label Phase: TMB-001 0.05% BID (N=38) | Maximal Use (N=34)
Application site dermatitis (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Application site erosion (General disorders) | 14 (18) | 2 (2) | 0 (0) | 4 (8) | 7 (7)
Application site erythema (General disorders) | 27 (39) | 4 (4) | 5 (7) | 6 (14) | 11 (16)
Application site oedema (General disorders) | 6 (7) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Application site pain (General disorders) | 23 (41) | 5 (6) | 4 (5) | 3 (10) | 13 (17)
Application site pruritus (General disorders) | 12 (14) | 0 (0) | 0 (0) | 5 (7) | 5 (7)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 3 (3) | 2 (3) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 7 (8) | 1 (3) | 0 (0) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT05295732/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT05295732/SAP_001.pdf